CLINICAL TRIAL: NCT02976857
Title: A Phase 1 Single Center, Non-randomized Study Evaluating Safety and Efficacy of Anti-CD19 Chimeric Antigen Receptor T-cell (C-CAR011) Treatment in Subjects With Refractory Diffuse Large B-cell Lymphoma
Brief Title: A Phase 1 Study Evaluating Safety and Efficacy of C-CAR011 Treatment in DLBCL Subjects
Acronym: C-CAR011
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai AbelZeta Ltd. (Industry)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBMG2016002
Record Dates: First submitted 2016-11-21; First posted 2016-11-29 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2016-11

CONDITIONS: Refractory Diffuse Large B-Cell Lymphoma
Keywords: refractory diffuse large B-cell lymphoma; anti-CD19 chimeric antigen receptor T-cell
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- C-CAR011 (Experimental): C-CAR011 infusion In the first cell therapy 0, 1 and 2 days, respectively 10%, 30% and 60% ratio three times reinfusion.
  Interventions: Biological: C-CAR-011

INTERVENTIONS:
Biological: C-CAR-011 — lymphocytes will be transduced with lentiviral vector containing CAR-CD19 gene.
  Other Names: CAR-CD19

SUMMARY:
The trial is a single arm, single-center, non-randomized phase I clinical trial which is designed to evaluate the safety and efficacy of C-CAR011 in treatment of refractory DLBCL

DETAILED DESCRIPTION:
The 3x3 dose escalation design will be adopted in order to determine the maximum tolerated dose (MTD). Subjects will be enrolled into low-dose group, medium-dose group and high-dose group as below:

Dose CAR+ cells/kg

Low 0.8×106

Medium 2.5×106

High 5.0×106

DLT is evaluated within 30 days post C-CAR011 infusion).

ELIGIBILITY:
Inclusion Criteria:

* Histologically diagnosed as DLBCL according to the NCCN non-Hodgkin's lymphoma Clinical Practice Guidelines (3rd edition 2016)
* Refractory DLBCL
* All subjects must have received adequate prior therapy including anti-CD20 monoclonal antibody (unless tumor is CD20-negative) and an anthracycline containing chemotherapy regimen. The standardized treatment regimens reference to NCCN non-Hodgkin lymphoma Clinical Practice Guidelines (2016 Version 3)
* At least one measurable lesion per revised IWG Response Criteria (the longest diameter of the tumor ≥ 1.5 cm)
* Age 18-70 years old, male or female
* Expected survival ≥ 12 weeks
* ECOG score 0-1
* Subject's left ventricular ejection fraction (LVEF) is ≥ 50% and no evidence of pericardial effusion as determined by an ECHO
* At least 4 weeks from receiving previous treatment (radiotherapy, chemotherapy, monoclonal antibody therapy or other treatments)
* No contraindications of peripheral blood apheresis
* Female subjects in childbearing age, their serum or urine pregnancy test must be negative, and must agree to take effective contraceptive measures during the trial measures
* Volunteered to participate in this study and signed informed consent

Exclusion Criteria:

* Have a history of allergy to cellular products
* Used any genetically modified T cell therapy
* History of allogeneic hematopoietic stem cell transplantation
* Severe active infection (uncomplicated urinary tract infections, bacterial pharyngitis allowed) or currently receiving intravenous antibiotic therapy and received intravenous antibiotic therapy within one week. Prophylactic antibiotic, antiviral and antifungal treatment is permissible
* Hepatitis B or hepatitis C virus infection (including carriers), as well as acquired, congenital immune deficiency diseases, including but not limited to HIV-infected persons
* Patients with class III and IV heart failure according to the NYHA Heart Failure Classifications
* A history of QT prolongation
* A history of epilepsy or other central nervous system disorders
* The patient had a history of other primary cancers, with the following exceptions: Excisional non-melanoma such as cutaneous basal cell carcinoma; Cured in situ carcinoma such as cervical cancer, bladder cancer or breast cancer
* Subjects with any autoimmune disease or any immune deficiency disease or other disease in need of immunosuppressive therapy
* Used of systemic steroids within two weeks (using inhaled steroids is an exception)
* Women who are pregnant or lactating or have breeding intent in 6 months
* Participated in any other clinical trial within three months
* The investigators believe that any increase in the risk of the subject or interference with the results of the trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-09-11 (Actual); Study Completion 2019-01-09 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 28 days
  Non-haematological dose-limiting toxicities was any toxicity of grade 3 or higher occurring within 28 days of C-CAR011 infusion judged possibly related to the treatment regimen.The following toxicities were not considered dose limiting toxicities: tumor lysis syndrome, abnormal electrolytes responding to supplementation, hypoalbuminemia, liver dysfunction resolving to ≤grade 2 within 14 days, transient (<72 hours) grade 4 hepatic enzyme abnormality, and grade 3 or 4 fever or neutropenic fever.

SECONDARY OUTCOMES:
Overall response rate | 4 and 12 weeks
  Overall response rate (ORR) = complete response (CR) rate + partial response (PR) rate, ORR will be assessed at weeks 4 and weeks 12 according to International Working Group (IWG) revised criteria.
Disease control rate | 12 weeks
  Disease control rate (DCR） = complete response (CR) rate + partial response (PR) rate + stable disease (SD) rate, DCR will be assessed at weeks 12 according to International Working Group (IWG) revised criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Jianyong Li, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Hematological Department, People's Hospital of Jiangsu Province, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338